CLINICAL TRIAL: NCT03327948
Title: Axonics SacRal NeuromodulaTIon System for Urinary Urgency Incontinence TreatmeNt (ARTISAN-SNM)
Brief Title: Axonics SacRal NeuromodulaTIon System for Urinary Urgency Incontinence TreatmeNt
Acronym: ARTISAN-SNM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105-0050
Record Dates: First submitted 2017-10-27; First posted 2017-11-01 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Urinary Incontinence, Urge
Keywords: Sacral neuromodulation (SNM); SNM
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment group (Experimental): Urinary Urgency Incontinence
  Interventions: Device: Axonics Sacral Neuromodulation System (SNM) System

INTERVENTIONS:
Device: Axonics Sacral Neuromodulation System (SNM) System — Axonics Sacral Neuromodulation System (SNM) System

SUMMARY:
The ARTISAN-SNM study is designed to evaluate the safety and effectiveness of the Axonics Sacral Neuromodulation System as an aid in the treatment of the symptoms of urinary urgency incontinence (UUI) in patients who have failed or could not tolerate more conservative treatments.

DETAILED DESCRIPTION:
The ARTISAN-SNM Trial which was a single-arm, prospective study that included 29 centers and enrolled 129 participants. The primary aim of the study was to evaluate the safety and efficacy of the Axonics SNM System for the treatment of UUI symptoms. Primary outcome was improvement in UUI episodes on a 3-day bladder diary. Secondary outcomes included quality of life using the ICIQ-OABqol questionnaire, patient satisfaction, and bowel symptoms captured using the Cleveland Clinic Florida Fecal Incontinence Score (CCF-FIS). Participants were followed out to 2 years and data was reported at 6 months, 1 year and 2 years

ELIGIBILITY:
Primary Inclusion Criteria:

1. Diagnosis of UUI demonstrated on a 72-hour voiding diary defined as a minimum of four (4) leaking episodes associated with urgency, at least 50% of all leaking episodes associated with urgency, and at least one leaking episode each 24-hour period.
2. Greater than or equal to 6 months' history of UUI diagnosis
3. For male subjects only: Peak flow rate > 15 cc/s as verified by uroflowmetry within 6 months prior to enrollment; Residual bladder volume < 150 cc tested within 6 months prior to enrollment
4. 21 years of age and older
5. Willing and capable of providing informed consent
6. Capable of participating in all testing associated with this clinical investigation

Primary Exclusion Criteria:

1. Stress incontinence or mixed incontinence.
2. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
3. Interstitial cystitis or bladder pain syndrome as defined by either American Urological Association (AUA) or European Association of Urology (EAU) guidelines
4. A female who is breastfeeding
5. A female with a positive urine pregnancy test

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Goldman, MD FACS, Principal Investigator — The Cleveland Clinic; Felicia Lane, MD, Principal Investigator — UC Irvine Health
Locations (4):
- United States (2):
  - UC Irvine Health, Irvine, California
  - Cleveland Clinic, Cleveland, Ohio
- Maastricht University Medical Center, Maastricht, Netherlands
- UCLH, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Group
Started | 129
Completed | 126
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 54
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [21 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 122
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 114
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Netherlands | 13
  United States | 97
  United Kingdom | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders
Description: Responders are defined as patients with greater than or equal to 50% reduction in symptoms
Time Frame: 2 years
Population: Completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 121
Participants | 113

2. Secondary Outcome: ICIQ-OAB-qol
Description: International Consultation on Incontinence Modular Questionnaire (ICIQ)- Overactive Bladder (OAB), Quality of Life (qol). Score range of 0-100, with greater values indicating better quality of life.
Time Frame: 2 years
Population: Completers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group
Number analyzed (Participants) | 121
score on a scale | 87.6 (13.9)

3. Secondary Outcome: Daily Number of Urgency Leaks
Description: The daily number of urgency leaks is measured by a bladder diary
Time Frame: 2 years
Population: Completers
Measure: Mean (Standard Deviation); unit: Daily number of UUI episodes
Arm/Group | Treatment Group
Number analyzed (Participants) | 121
Daily number of UUI episodes | 1.0 (1.7)

4. Secondary Outcome: Voids
Description: Measured by a bladder diary
Time Frame: 2 years
Population: Completers
Measure: Mean (Standard Error); unit: Voids
Arm/Group | Treatment Group
Number analyzed (Participants) | 121
Voids | 8.5 (2.4)

5. Other Pre Specified Outcome: Change in CCF-FIS Score for Participants With a CCF-FIS Score ≥6 at Baseline
Description: Change in CCF-FIS score at follow-up compared to baseline. Cleveland Clinic Florida - Fecal Incontinence Score (CCF-FIS): includes 5 items (solid, liquid, gas, wears pad and lifestyle alteration) and 5 frequencies (never = 0, rarely = 1, sometimes = 2, usually = 3, always = 4). Scores range from 0 for full continence to 20 for complete incontinence. A higher score indicates more severe FI symptoms and a score ≥ 6 indicates moderate to severe FI symptoms.
Time Frame: Baseline, 2-years
Population: Completers
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Fecal Incontinence: Subjects with a score of ≥6 at baseline were determined to have fecal incontinence
Arm/Group | Fecal Incontinence
Number analyzed (Participants) | 42
score on a scale
  Baseline | 9.3 (3.3)
  2-years | 3.7 (3.4)

6. Other Pre Specified Outcome: Participant Satisfaction for Treatment of UUI Symptoms
Description: The subject satisfaction questionnaire was designed to provide information on subjective satisfaction with r-SNM therapy and the recharging experience. Participants indicated satisfaction with r-SNM therapy for treatment of their UUI symptoms based on a 7-point Likert scale ranging from "Very satisfied" to "Very dissatisfied". Results are presented as the number of participants who reported "Very, moderately, or slightly satisfied" with r-SNM therapy for treatment of their UUI symptoms.
Time Frame: 2-year
Population: Completers
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 121
Participants | 114

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 1/129
Serious Adverse Events (participants affected / at risk) | 19/129
Other Adverse Events (participants affected / at risk) | 20/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=129)
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Appendicitis (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Influenza like illness (General disorders) | 1
Bilary sepsis (Infections and infestations) | 1
Chlostridium difficile infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Incision site infection (Infections and infestations) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthalgia (Musculoskeletal and connective tissue disorders) | 1
Paresis (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=129)
Proctalgia (Gastrointestinal disorders) | 1
Implant site coldness (General disorders) | 1
Medical device site pain (General disorders) | 1
Medical device discomfort (General disorders) | 2
Implant site pain (General disorders) | 3
Incision site infection (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Paraesthesia (Nervous system disorders) | 1
Lead dislodgement (Product Issues) | 1
Device power source issue (Product Issues) | 3
Device breakage (Product Issues) | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1
Medical device change (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03327948/Prot_SAP_000.pdf